CLINICAL TRIAL: NCT04604665
Title: Evaluation of the Efficacy of Two Levels of Frequency of Repositioning in Adults Hospitalized in Intensive Care Units, in the Reduction of Pressure Ulcers: A Randomized Cluster Study.
Brief Title: Evaluation of Two Levels of Frequency of Repositioning in the Reduction of Pressure Ulcers
Acronym: PENFUP-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Cardioinfantil Instituto de Cardiología (Other)
Collaborators: Universidad Autónoma de Bucaramanga (Other)
Responsible Party: Principal Investigator, Olga Cortés, RN, MSc, PhD, Reseear Associated, Research Department, Principal Investigator, Fundación Cardioinfantil Instituto de Cardiología
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 844-2019
Record Dates: First submitted 2020-10-14; First posted 2020-10-27 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Clinical trial, randomized, pragmatic, of parallel groups (1: 1), by clusters, blinded for the collection of information, sending, and in the evaluation of outcomes.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Telephone randomization Random numbers centers Blinded for analyst and researchers
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High frequency postural change (Experimental): Repositioning or rotation of patients hospitalized in bed in intensive care units will be carried out with a frequency interval that we call "high-frequency". It has to be performed on each patient between an interval less than or equal to every 2 hours in a full day (24 hours) (minimum goal of 8-10 in 24 hours subtracting 2 or 4 at night and not alter the circadian cycle). The position must be modified in each postural change to the right lateral, supine, left lateral, supine, or prone position to supine position. The repositioning will be provided until a patient is discharged from ICU, die or begin ambulation. When providing each repositioning, avoid dragging the patient, the shear, and the friction to increase UPP risk. This must be applied to avoiding massage. Patients in any position should use pressure-reducing items such as pillows.
  Interventions: Other: High frequency postural change
- Conventional care (Active Comparator): Repositioning or rotation of patients hospitalized will be the conventional or usual care. Units in this group are not going to receive any intervention. Will be only observed in their current intervention of repositioning.
  Interventions: Other: Conventional care

INTERVENTIONS:
Other: High frequency postural change — Repositioning of patients hospitalized in bed in intensive care units will be carried out with a frequency interval that we call "high-frequency" to be performed on each patient between an interval between less than or equal to every 2 hours in a full day (24 hours) (minimum goal of 8-10 in 24 hours subtracting 2 or 4 at night and not alter the circadian cycle). The position must be modified in each postural change to right lateral, supine, left lateral, or prone to supine if the position changes every 2 hrs.
  Other Names: Repositioning
  Arms: High frequency postural change
Other: Conventional care — Repositioning of patients hospitalized will be performed in the current way it is commonly applied to patients.
  Other Names: Control group or usual or current care
  Arms: Conventional care

SUMMARY:
PENFUP FASE 2, It is a multicenter study by parallel conglomerates, planned in order to evaluate the efficacy between two levels of frequency of postural change in intensive care units for adults of hospitals in various regions of Colombia.

DETAILED DESCRIPTION:
Taking into account a design effect of 6.7, Investigators planned to include 150 participants from each ICU. Investigators did calculate that a total of 22 ICUs are required, in which 11 will be assigned to the low frequency and 11 will be assigned to a high frequency group of postural change until obtaining a total of 1,650 patients in each arm of the study and a total of 3,300 participants in the study.

ELIGIBILITY:
Inclusion Criteria:

* The ICU manage adult patients, over 18 years of age, with any type of emphasis (surgical, medical, neurological, or mixed);
* Patients are admitted in critical condition (with life support);
* The director accepts the commitment of the care assigned in the randomization (for a period of 3 months).

Exclusion Criteria:

* Intermediate care units in which patients mobilize themselves.
* Covid patients or other patients exposed to different mobilization patterns (e.g., 12 hours prone vs 12 supine)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3300 (Actual)
Dates: Start 2021-04-10 (Actual); Primary Completion 2023-12-10 (Actual); Study Completion 2023-12-10 (Actual)

PRIMARY OUTCOMES:
The incidence (incidence rata ration) of new pressure ulcers in each Intensive Care Unit (ICU) | " 1 month after admission"
  The number of pressure injuries at any stage, new acquired in the ICU after admission per 1,000 patient days in the ICU.

SECONDARY OUTCOMES:
Risk index (HR) and time to event of Pressure ulcers of the patients | "1 month safter admission"
  Hazard ratio and tiem to event of PUs of patients included in the repositioning group with the lowest frequency compared to the group of patients included by intervention group in the development of the first PU during their stay in the ICU.
Security outcomes | "1 month after admission"
  Secondary safety outcomes: includes possible complications associated with postural changes: permanent or sporadic changes in ventilatory parameters (hypoxemia), hemodynamic changes (tachycardia, hypertension); events such as acute respiratory failure; or cardiogenic shock, pneumonia.

CONTACTS AND LOCATIONS:
Overall Officials: Olga L Cortés, PhD, Principal Investigator — Fundación Cardioinfantil Instituto de Cardiología
Locations (21):
- Colombia (21):
  - Hospital IPS Universitaria, Medellín, Antioquia
  - Hospital San Vicente de Paul, Medellín, Antioquia
  - Hospital San Vicente_RioNegro, Rionegro, Antioquia
  - Hospital Central Barranquilla, Barranquilla, Atlántico
  - Clínica Palermo, Bogotá, Bogota D.C.
  - Hospital Militar Central, Bogotá, Bogota D.C.
  - Hospital San José, Bogotá, Bogota D.C.
  - S.E.S Hospital Universitario de Caldas, Manizales, Caldas Department
  - Centro Policlínico de Olaya, Bogotá, Cundinamarca
  - Clinica Nogales, Bogotá, Cundinamarca
  - Fundación CardioInfantil Instituto de Cardiología, Bogotá, Cundinamarca
  - Hospital Erasmo Meoz, Cúcuta, Norte de Santander Department
  - Fundación Cardiovascular Bucaramanga, Bucaramanga, Santander Department
  - International Hospital of Colombia -HIC, Bucaramanga, Santander Department
  - Hospital Federico Lleras Acosta, Ibagué, Tolima Department
  - Hospital Universitario Norte Barranquilla, Barranquilla
  - Clínica de Occidente, Bogotá
  - Clínica SHAIO, Bogotá
  - Hospital Universitario La Samaritana, Bogotá
  - Clìnica FOSCAL Internacional, Bucaramanga
  - Clìnica Foscal_Carlos Ardila lulle, Bucaramanga

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gillespie BM, Chaboyer WP, McInnes E, Kent B, Whitty JA, Thalib L. Repositioning for pressure ulcer prevention in adults. Cochrane Database Syst Rev. 2014 Apr 3;2014(4):CD009958. doi: 10.1002/14651858.CD009958.pub2. PMID 24700291
- [Background] Ulrika Källman. (2015). Evaluation of Repositioning in Pressure Ulcer Prevention. Linköping University Medical Dissertations No. 1455. Division of Nursing science Department of Medical and Health Sciences. Linköping University, Sweden.
- [Background] Hawkins S, Stone K, Plummer L. An holistic approach to turning patients. Nurs Stand. 1999 Oct 6-12;14(3):51-6. doi: 10.7748/ns1999.10.14.3.51.c2689. PMID 10983058
- [Background] Burk RS, Grap MJ. Backrest position in prevention of pressure ulcers and ventilator-associated pneumonia: conflicting recommendations. Heart Lung. 2012 Nov-Dec;41(6):536-45. doi: 10.1016/j.hrtlng.2012.05.008. Epub 2012 Jul 21. PMID 22819601
- [Background] Eldridge S., Kerry S. Designing interventions in: A practical guide to cluster randomized trials in health services research. Page 44-57. Centre for Primary Care and Public Health, Barts, and The London School of Medicine and Dentistry, Queen Mary University of London UK. 2012 John Wiley & Sons, Ltda.
- [Derived] Cortes OL, Herrera-Galindo M, Villar JC, Rojas YA, Del Pilar Paipa M, Salazar L. Frequency of repositioning for preventing pressure ulcers in patients hospitalized in ICU: protocol of a cluster randomized controlled trial. BMC Nurs. 2021 Jul 5;20(1):121. doi: 10.1186/s12912-021-00616-0. PMID 34225724